CLINICAL TRIAL: NCT05823376
Title: Efficacy and Safety of Avatrombopag for Platelet Recovery After Unrelated Cord Blood Transplantation in Patients With Bone Marrow Failure Disease: a Single-center, Single-arm, Phase II Trial
Brief Title: Avatrombopag for Platelet Recovery Post-UCBT in Patients With Bone Marrow Failure Disease
Acronym: AVA
Status: Recruiting | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Xiaoyu Zhu, Chief physician, Anhui Provincial Hospital
Other Study IDs: AVA&MDS-001
Record Dates: First submitted 2023-03-24; First posted 2023-04-21 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Platelet Recovery After Umbilical Cord Blood Transplantation
Keywords: Avatrobopag
MeSH Terms: interventions — avatrombopag

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Avatrombopag group: The duration of the study is 4 weeks, from +1 day to +28 days after UCBT, patients will be given Avatrombopag with a recommended dose of 40mg per day. After 28 days of administration, the patients may continue, change or discontinue medication based on the patients' platelet status.
  Interventions: Drug: Avatrombopag

INTERVENTIONS:
Drug: Avatrombopag — Indications for drug reduction and withdrawal: excluding blood transfusion factors, the reduction will be 20mg/d when PLT≥50×10^9/L; Drug administration will be stopped when PLT≥100×10^9/L.

SUMMARY:
To evaluate the efficacy and safety of Avatrombopag for platelet recovery after unrelated cord blood transplantation (UCBT) in patients with bone marrow failure disease

DETAILED DESCRIPTION:
Persistent thrombocytopenia is a common complication after umbilical cord blood transplantation (UCBT), which necessitates platelet transfusion and leads to increased transplant-related mortality. This is a single-center, single-arm, phase II clinical trial aimed at evaluating the efficacy and safety of Avatrombopag for platelet recovery after UCBT in patients with bone marrow failure disease (BMFD). The study was conducted in patients diagnosed with BFMD and receiving UCBT. After the subjects signed and informed and qualified, they received Avatrombopag treatment from the first day to the 28th day after transplantation. In this study, the cumulative of platelet implantation rate at 28 days after transplantation was used as the main therapeutic index, and 40 patients were planned to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥12 years old, male or female;
* Patients diagnosed with bone marrow failure disease including aplastic anemia (AA), Fanconi anemia (FA), paroxysmal nocturnal hemoglobinuria (PNH) and undergoing UCBT;
* ECOG score ≤2;
* Voluntary participation in this clinical trial, patients fully understand the trial content and sign the informed consent；

Exclusion Criteria:

* Pregnant or lactating women；
* Known allergy to Avatrombopag;
* A history of severe thrombotic events or known risk factors for thrombosis or active thromboembolism requiring anticoagulation;
* A history of platelet dysfunction or bleeding prone disease or severe bleeding (requiring more than 2 units of red blood cell infusion or a hematocrit drop of ≥10%) within 7 days prior to screening;
* Chronic active hepatitis B and C;
* Repeat or multiple transplantation or multiple organ transplantation;
* HIV positive, EBV-DNA positive, CMV-DNA positive;
* Have severe infection or complicated with serious heart, liver, lung, kidney, neurological or metabolic diseases;
* A serious adverse event (Level 4 or 5) as defined by the Standard General Terminology for Adverse Events Version 4.0 occurred during the pre-treatment period;
* Participants participate in another clinical study with any exploratory drug or device within 30 days prior to baseline visit; Observational studies are allowed;
* Subjects with cognitive impairment or uncontrolled mental illness;
* Subjects and/or authorized family members to refuse treatment with Avatrombopag;
* Those who are judged by the researchers as not suitable for inclusion (such as accompanying medical history, which may affect the safety of the subjects or it is estimated that the treatment cannot be adhered to due to financial problems).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with bone marrow failure and receiving umbilical cord blood transplantation
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Time of platelet engraftment | 28 days
  Platelet engraftment is defined as independence from platelet transfusion for at least 7 days with a platelet count of more than ≥20 × 10^9/L.
The cumulative incidence of platelet engraftment at 28 days after transplantation | 28 days
  Platelet engraftment is defined as independence from platelet transfusion for at least 7 days with a platelet count of more than ≥20 × 10^9/L.

SECONDARY OUTCOMES:
The cumulative incidence of platelet recovery rate at 28 days after transplantation | 28 days
  Platelet recovery was defined as independence from platelet transfusion for at least 7 days with a platelet count of more than ≥50×10^9/L.
Total platelet transfusion during 4 weeks of treatment | 28 days
  Total platelet transfusion during 4 weeks of treatment
neutrophil reconstitution | 28 days
  neutrophil engraftment time was defined as the first of three consecutive days during which the neutrophil count was at least 0.5×10^9/L.
erythroid reconstitution | 28 days
  RBC engraftment time was defined as the first day of achieving a reticulocyte count greater than 1% for 3 consecutive days.
Megakaryocyte levels in bone marrow smears 4 weeks after treatment | 4 weeks
  Megakaryocyte levels in bone marrow smears 4 weeks after treatment
Time of platelet recovery | 100 days
  Platelet count ≥50×10^9/L for 3 consecutive days without platelet transfusions for 7 consecutive days
Time of platelet ≥100×10^9/L. | 100 days
  Platelet count ≥100×10^9/L for 3 consecutive days without platelet transfusions for 7 consecutive days

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyu Zhu, ph.D, Principal Investigator — The First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital)
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital), Hefei, Anhui, China